CLINICAL TRIAL: NCT05519696
Title: The Together Everyone Achieves More Physical Activity Trial
Brief Title: Together Everyone Achieves More (TEAM) Trial
Acronym: TEAM
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of South Carolina (Other)
Collaborators: National Heart, Lung, and Blood Institute (NHLBI) (NIH)
Responsible Party: Principal Investigator, Allison M. Sweeney, Assistant Professor, University of South Carolina
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: Pro00113152; R01HL160618 (NIH)
Record Dates: First submitted 2022-08-22; First posted 2022-08-29 (Actual); Last update posted 2024-10-24 (Actual); Status verified 2024-10

CONDITIONS: Physical Activity
Keywords: African American women; Community-Based Intervention; Social Environment
MeSH Terms: conditions — Motor Activity | interventions — Methods

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: All measurement staff will be blind to treatment condition
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): This group will receive a 10-week group-based intervention program.
  Interventions: Behavioral: Intervention
- Comparison (Active Comparator): The group will receive a 10-week group-based comparison program.
  Interventions: Behavioral: Comparison

INTERVENTIONS:
Behavioral: Intervention — Participants receiving the intervention will complete a 10-week group program. Group sessions meet once per week for 2 hours and include three components - discussion-based health promotion initiative, team-based physical activity games/activities, and team-based goal-setting and behavioral skills training. The health promotion initiative uses cultural targeting and includes a focus on cultural topics related to collectivism. Participants receive FitBits to track their physical activity and through the FitBit mobile app are connected to their group members to encourage communication and social support.
  Arms: Intervention
Behavioral: Comparison — Participants receiving the comparison program will complete a 10-week group program. Group sessions meet once per week for 2 hours and include three components - discussion-based health promotion initiative, group walking program, and individual-based goal-setting and behavioral skills training. The health promotion initiative uses cultural targeting only (and no focus on collectivism). Participants receive FitBits to track their physical activity, but are not connected to their group members on the mobile app.
  Arms: Comparison

SUMMARY:
The Together Everyone Achieve More (TEAM) Physical Activity trial evaluates the efficacy of a group-based social affiliation intervention (vs. a standard group-delivered physical activity comparison program) for increasing physical activity among inactive African American women. Using a group cohort randomized design implemented at community centers across five years, the primary aim of this study is to evaluate the efficacy of the 10-week TEAM-PA group-based intervention (vs. comparison program) on increasing daily total physical activity from baseline to post-intervention and maintenance at a 6-month follow-up.

ELIGIBILITY:
Inclusion Criteria:

* at least 18 years of age
* self-identifying as an African American or Black female
* engaging in < 60 minutes of moderate to vigorous physical activity per week for the last three months

Exclusion Criteria:

* having a cardiovascular or orthopedic condition that would limit physical activity (including walking with a cane/walker)
* currently pregnant or planning to become pregnant in the next 2 months
* uncontrolled blood pressure (systolic >180 mmHg/diastolic > 110 mmHg)

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 360 (Estimated)
Dates: Start 2022-09-12 (Actual); Primary Completion 2026-12 (Estimated); Study Completion 2026-12 (Estimated)

PRIMARY OUTCOMES:
Total Physical Activity | Baseline, post-intervention (10 weeks), and 6 months post-intervention
  Average minutes of total physical activity (PA) per day; Objective assessments of total PA will be obtained with ActiGraph accelerometers. Participants will wear the monitor on the non-dominant wrist for 7 consecutive days. The investigators will evaluate whether there is a change in minutes of total PA per day from baseline to 10 weeks and maintenance at 6 months post-intervention, and whether there are group differences between the intervention and comparison programs.

SECONDARY OUTCOMES:
Percentage meeting national guidelines for weekly moderate to vigorous physical activity | Baseline, post-intervention (10 weeks), and 6 months post-intervention
  Percentage of participants with at least 150 minutes of moderate physical activity and/or 75 minutes of vigorous physical activity per week; Objective assessments of minutes of moderate to vigorous physical activity will be obtained with ActiGraph accelerometers. The investigators will evaluate whether there is a change in the percentage of participants meeting national guidelines from baseline to 10 weeks and maintenance at 6 months post-intervention, and whether there are group differences between the intervention and comparison programs.
Light Physical Activity | Baseline, post-intervention (10 weeks), and 6 months post-intervention
  Average minutes of light physical activity (PA) per day; Objective assessments of light PA will be obtained with ActiGraph accelerometers. The investigators will evaluate whether there is a change in daily minutes of light PA from baseline to 10 weeks and maintenance at 6 months post-intervention, and whether there are group differences between the intervention and comparison programs.
Sedentary Behavior | Baseline, post-intervention (10 weeks), and 6 months post-intervention
  Average minutes of sedentary behavior per day; Objective assessments of sedentary behavior will be obtained with ActiGraph accelerometers. The investigators will evaluate whether there is a change in sedentary behavior from baseline to 10 weeks and maintenance at 6 months post-intervention, and whether there are group differences between the intervention and comparison programs.
Body Mass Index (BMI) | Baseline, post-intervention (10 weeks), and 6 months post-intervention
  Height (cm) and weight (kg) will be measured using a stadiometer and medical-grade scale. Scores will be used to calculate BMI (kg/m^2). The investigators will evaluate whether there is a change in BMI from baseline to 10 weeks and maintenance at 6 months post-intervention, and whether there are group differences between the intervention and comparison programs.
Blood Pressure | Baseline, post-intervention (10 weeks), and 6 months post-intervention
  Systolic and diastolic blood pressure will be measured using an automatic blood pressure machine. The investigators will evaluate whether there is a change in blood pressure from baseline to 10 weeks and maintenance at 6 months post-intervention, and whether there are group differences between the intervention and comparison programs.
Two-Minute Walk Test (Walking Speed) | Baseline, post-intervention (10 weeks), and 6 months post-intervention
  Starting from a standing position, participants are asked to walk as far as they can in a safe manner for two minutes over a flat out and back 50 feet course. The distance traveled to the nearest foot is recorded.

OTHER OUTCOMES:
Reciprocal Social Support for Physical Activity | Baseline, post-intervention (10 weeks), and 6 months post-intervention
  The Support for Exercise Scale (Sallis et al 1987) will be adapted [12 items; 1 = Never; 6 = Very Frequently ] to measure providing and receiving of social support among group members. Mean composite scores will be calculated (ranging from 1-6), with higher numbers indicate greater social support.
Group Cohesion among Group Members | Baseline, post-intervention (10 weeks), and 6 months post-intervention
  Two subscales (Individual Attraction to the Group - Social; Group Integration - Social) from the Physical Activity Group Environment Questionnaire (Estrabrooks et al 2000) [10 items; 1 = Strongly Disagree, 6= Strongly Agree] will be used to assess group cohesion among group members. Mean composite scores will be calculated (ranging from 1-6), with higher numbers indicate greater group cohesion.
Group Interactions (Communication, Cooperation, Friendly Competition) | Baseline, post-intervention (10 weeks), and 6 months post-intervention
  Items developed by Harden et al (2014) [12 items; 1 = Strongly Disagree, 6= Strongly Agree] will be used to assess communication, cooperation, and friendly competition among group members. Mean composite scores will be calculated (ranging from 1-6), with higher numbers indicate more positive group interactions.
Collective Efficacy for Physical Activity among Group Members | Baseline, post-intervention (10 weeks), and 6 months post-intervention
  The Unity subscale from the Collective Efficacy Questionnaire for Sports (Short et al. 2005) will be adapted [4 items; 5-point, 1 = Not at all confident, 5 = Extremely confident] to assess collective efficacy for physical activity among group members. A mean composite score will be calculated (ranging from 1-5), with higher numbers indicating greater collective efficacy.
Relatedness among Group Members | Baseline, post-intervention (10 weeks), and 6 months post-intervention
  The Need for Relatedness Scale (Richer & Vallerand, 1998) will be used [10 items; 1 = Strongly Disagree, 6= Strongly Agree] to assess relatedness among group members. A mean composite score will be calculated (ranging from 1-6), with higher numbers indicating greater relatedness.

CONTACTS AND LOCATIONS:
Locations (1):
- College of Nursing, University of South Carolina, Columbia, South Carolina, United States

IPD SHARING:
Plan to Share IPD: No
The investigators plan to share the Statistical Analysis Plan and Informed Consent Form.

REFERENCES:
- [Derived] Sweeney AM, Wilson DK, Zarrett N, Simmons T, Mansfield M, Decker L. Using formative process evaluation to improve program implementation and accessibility of competitive group-based physical activity in the TEAM-PA trial. Int J Behav Nutr Phys Act. 2024 Aug 13;21(1):88. doi: 10.1186/s12966-024-01635-1. PMID 39138496
- [Derived] Sweeney AM, Wilson DK, Zarrett N, Martin P, Hardin JW, Fairchild A, Mitchell S, Decker L. An overview of the Together Everyone Achieves More Physical Activity (TEAM-PA) trial to increase physical activity among African American women. Contemp Clin Trials. 2023 Jun;129:107207. doi: 10.1016/j.cct.2023.107207. Epub 2023 Apr 26. PMID 37116644